CLINICAL TRIAL: NCT04866706
Title: Performance and Safety of Routine Cataract Surgery With Visiol
Status: Completed | Type: Observational
Sponsor: TRB Chemedica (Industry)
Responsible Party: Sponsor
Other Study IDs: SVS18-CT-1901
Record Dates: First submitted 2021-04-18; First posted 2021-04-30 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-04

CONDITIONS: Following Cataract Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Visiol — VISIOL is a 2.0% (m/v) SH viscoelastic solution used for ocular surgery.
  Other Names: Sodium hyaluronate

SUMMARY:
In this clinical investigation, the performance and safety of routine cataract surgery with VISIOL will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years and older;
* Candidate for cataract surgery via phacoemulsification;
* Ophthalmic surgeon's recommendation to use VISIOL prior to recruitment;
* Eligible for the use of VISIOL as indicated in the instructions for use;
* Written informed consent.

Exclusion Criteria:

* Known allergy or hypersensitivity to any of VISIOL components;
* Known pregnancy or breast feeding;
* Participation in any other clinical research study within the last 90 days;
* Patients with legally restricted autonomy, freedom of decision and action (e.g. those with measure of custody or judicial protection);
* Incapacity to understand the informed consent and/or to comply with the Clinical Investigation Plan (CIP), per investigator's appreciation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over 18 years cataract patients whom investigator routine considered to treat by surgery with Visiol before recruit to study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Corneal endothelial cells density in percent | Change from pre-surgery Corneal endothelial cells density at Day 1, Day 7, Day 30, Day 90
  The variation of corneal endothelial cells density (cells/mm2) as compared to baseline (pre-surgery) will be calculated (%)

OTHER OUTCOMES:
Corneal endothelial cells area | Change from pre-surgery Corneal endothelial cells area at Day 1, Day 7, Day 30, Day 90
  The area (µm2) of corneal endothelial cells will be measured using a non-contact specular microscopy.
Corneal endothelial cells density | Change from pre-surgery Corneal endothelial cells density at Day 1, Day 7, Day 30, Day 90
  The density (cells/mm2) of corneal endothelial cells will be measured using a non-contact specular microscopy.
Corneal endothelial cells regularity | Change from pre-surgery Corneal endothelial cells regularity at Day 1, Day 7, Day 30, Day 90
  The regularity (variation of size) of corneal endothelial cells will be measured using a non-contact specular microscopy. In particular, the endothelial regularity will be assessed using the following classification described in ISO 11980:2012:37 0 = Regular endothelial mosaic;
  1. = Isolated difference in cell size;
  2. = Just noticeable variation in cell size or bumpiness of cell layer;
  3. = Easily detected difference in cell size or bumpiness of cell layer;
  4. = Noticeable cell layer bumpiness and loss of definition of cell borders.
The presence of keratic precipitates | Change from pre-surgery presence of keratic precipitate at Day 1, Day 7, Day 30, Day 90
  The presence (0 = No, 1 = Yes) of Keratic precipitate will be recorded
A description of keratic precipitates type | Change from pre-surgery a description of keratic precipitates type at Day 1, Day 7, Day 30, Day 90
  A description of keratic precipitates type will be recorded
Central corneal thickness | Change from pre-surgery central corneal thickness at Day 1, Day 7, Day 30, Day 90
  Central corneal thickness (micrometer) will be measured using non-contact specular microscopy
Corneal oedema | Change from pre-surgery corneal oedema at Day 1, Day 7, Day 30, Day 90
  Corneal oedema grading will be assessed using a specular microscopy. Gradings will be referred to location of oedema
  1. = Peripheral oedema
  2. = Central oedema
  3. = Generalised oedema
Intra-ocular pressure | Change from pre-surgery intra-ocular pressure at Day 0 (surgery day), Day 1, Day 7, Day 30, Day 90
  Intra-ocular pressure (mmHg) will be evaluated using a Goldmann applanation tonometry
Incidence of intra-ocular pressure peak | Change from pre-surgery intra-ocular pressure peaks at Day 0 (surgery day), Day 1, Day 7, Day 30, Day 90
  The incidence of intra-ocular pressure peaks (≥ 30 mmHg) will be recorded
Anterior chamber inflammation cell | Change from pre-surgery anterior chamber inflammation cell at Day 1, Day 7, Day 30, Day 90
  Anterior chamber inflammation will be assessed using slit lamp biomicroscopy (1 mm slit beam). It will be classified based on SUN grading Grade 0 = < 1 cell in field Grade 0.5 = 1-5 cells in field Grade 1 = 6-15 cells in field Grade 2 = 16-25 cells in field Grade 3 = 26-50 cells in field Grade 4 = over 50 cells in field
Anterior chamber inflammation flare | Change from pre-surgery anterior chamber inflammation flare at Day 1, Day 7, Day 30, Day 90
  Anterior chamber inflammation will be assessed using slit lamp biomicroscopy (1 mm slit beam). It will be classified based on SUN grading Grade 0 = no flare Grade 1 = faint Grade 2 = moderate (iris/ lens details clear) Grade 3 = marked (iris/ lens details hazy) Grade 4 = Intense (fibrin/ plastic aqueous)
Best corrected visual acuity (BCVA) | Change from pre-surgery BCVA at Day 1, Day 7, Day 30, Day 90
  BCVA will be evaluated using standard ETDRS logMAR chart
Intra-surgery information for duration of intervention | During Surgery (Day 0)
  duration of intervention (min)
Intra-surgery information for use of finger grip | During Surgery (Day 0)
  Use of finger grip (yes or no)
Intra-surgery information for time needed to remove VISIOL | During Surgery (Day 0)
  Time needed to remove VISIOL (min) counted from the time when intra-ocular lens was inserted until when the aspiration tip is removed
Intra-surgery information for volume of VISIOL used | During Surgery (Day 0)
  Total volume of VISIOL used (mL)
Intra-surgery information for material of intra-ocular lens used | During Surgery (Day 0)
  Material of intra-ocular lens used (acrylic or silicone)
Intra-surgery information for power of intra-ocular lens used | During Surgery (Day 0)
  Power (diopters) of intra-ocular lens used
Intra-surgery information for incision size | During Surgery (Day 0)
  Incision size (mm)
Intra-surgery information for energetic parameter power or energy | During Surgery (Day 0)
  Power or energy (% or mJ) during phacoemulsification and photolysis
Intra-surgery information for time of phacoemulsification | During Surgery (Day 0)
  Time (min) during phacoemulsification
Intra-surgery information for vacuum | During Surgery (Day 0)
  Vacuum (mmHg) during phacoemulsification
Investigator's subjective judgement | During Surgery (Day 0)
  using a 4 point grading scale: ease of VISIOL injection, maintenance of the anterior chamber depth during the capsulorhexis and IOL implantation, ability to remain in the anterior chamber during phacoemulsification and photolysis, clarity of the substance, ease of capsulorhexis, ease of IOL implementation, ease of VISIOL removal and global impression on the product performance during the surgery. Grading scale will be assessed 0 = Not effective
  1. = slightly effective
  2. = moderately effective
  3. = very effective
Global evaluation of the performance by the investigator | Surgery day (Day 0) and Day 90
  Global evaluation of the performance of cataract surgery with VISIOL by the investigator 0 = no improvement
  1. = slight improvement
  2. = moderate improvement
  3. = great improvement
Global evaluation of the performance by the patient | Surgery day (Day 0) and Day 90
  Global evaluation of the performance of cataract surgery with VISIOL by the patient 0 = no improvement
  1. = slight improvement
  2. = moderate improvement
  3. = great improvement
Adverse events (AE) | Pre-surgery, Surgery day (Day 0), Day 1, Day 7, Day 30, Day 90
  including their incidence, intensity, seriousness, expectedness and causal relationship with the use of investigational device or study procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand